CLINICAL TRIAL: NCT01688219
Title: Immune Mechanisms During SAPHO Syndrome and Treatment by Etarnecept
Brief Title: Immune Response in the SAPHO Syndrome
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 45896566645469
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2007-10

CONDITIONS: SAPHO Syndrome
Keywords: SAPHO syndrome; Innate immunity; TNF alpha; Polymorphonuclear neutrophils; Propionibacterium acnes; Interleukin-8
MeSH Terms: conditions — Acquired Hyperostosis Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aetiology of SAPHO syndrome seems to involve genetic, infectious and immunological components. The investigators examined innate and adaptative immune responses in SAPHO syndrome as compared with psoriatic arthritis and rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SAPHO syndrome
* Must have bone lesions

Exclusion Criteria:

* Infliximab treatment

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: SAPHO syndrome patients
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2005-11; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
IL-8 production by PMN | 24 h

SECONDARY OUTCOMES:
TNFalpha production by PMN | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Hayem, PhD, Study Director — Assitance Publique-Hopitaux Paris